CLINICAL TRIAL: NCT05722223
Title: Trimodal Prehabilitation in Pancreatic Cancer Patients Candidate to Neoadjuvant Treatment: A Pilot Study
Brief Title: Trimodal Prehabilitation in Pancreatic Cancer Patients Urdergoing Neoadjuvant Treatment
Acronym: PREPANC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Ana Ruiz-Casado, Medical oncologist, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PH-UMH02
Record Dates: First submitted 2022-03-14; First posted 2023-02-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Neoplasms
Keywords: exercise; pancreatic; cancer; trimodal
MeSH Terms: conditions — Pancreatic Neoplasms; Motor Activity; Neoplasms

STUDY DESIGN:
Intervention Model Description: All the participants will receive trimodal prehabilitation. Only one arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training group (Experimental): Pancreatic patients will participate in the trimodal prehabilitation: nutrition, psychological and exercise support.
  Interventions: Combination Product: Trimodal prehabilitation

INTERVENTIONS:
Combination Product: Trimodal prehabilitation — Pancreatic cancer patients (not stage 4) will undergo trimodal prehabilitation: nutrition, psychological, and exercise support.

SUMMARY:
Pancreatic cancer is a disease with a very poor prognosis and less than 10% of these patients live beyond 5 years from diagnosis. Further, it is expected to become the second leading cause of death in the coming years. Today, surgery remains the cornerstone in curing this disease, but the addition of chemotherapy is needed to improve survival. The impact of adjuvant treatment has been previously demonstrated and its efficacy is absolute. However, neoadjuvant chemotherapy (pre-surgery) improves the results after surgery (achieving earlier stages and with better prognosis) and would lead to better survival results. Besides, the moment of cancer diagnosis is a moment of special receptivity to change lifestyles ("teachable moment").

Multimodal prehabilitation includes 1) physical exercise; 2) nutritional and 3) psychological support. The potential advantages of prehabilitation during neoadjuvant therapy would be 1) the possibility of achieving a better physical condition to face surgery; 2) fewer postoperative complications; 3) more likely to receive adjuvant treatment after surgery; 4) better physical function at the end of treatments. To date, most studies have focused on lung and prostate cancer, with a high prevalence of men in the series.

This strategy has previously been explored, showing that it is safe and feasible, (Loughney et al). We have not identified any study of trimodal prehabilitation during neoadjuvant treatment and none that has integrated motivational strategies to maintain adherence.

Patients during chemotherapy have perceived several adverse effects that could limit adherence to the program. In this regard, a review on the motivation and exercise in cancer survivors shows that it is necessary to apply theoretical frameworks to understand cognitive and motivational processes and develop educational interventions. The self-determination theory is one of the motivational theories most applied today to the analysis of factors related to the adoption of healthy lifestyles. Likewise, patients who are motivated are more likely to improve healthy habits and obtain greater adherence to exercise performance. Therefore, we aimed of carrying out an intervention (pilot study) in ten patients to describe the feasibility of a trimodal prehabilitation program in the hospital environment, applying motivational strategies and a mixed-method (face-to-face and online).

DETAILED DESCRIPTION:
outcome measures refer to feasibility of the intervention:

Recruitment Attendance to the training sessions Attendance to psychologist and nutritionist sessions

And also to physical condition Cardiorespiratory fitness Muscular strength Body composition Physical activity Quality of life Fatigue score

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* ECOG 0-2
* Being able to complete the mile-time test
* Stages I-III
* Being able to understand the informed consent
* Pancreatic cancer diagnosed

Exclusion Criteria:

* Metastasic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
To explore the feasibility of a trimodal prehabilitation program in the hospital setting | 1 year
  Adherence to 70% of supervised physical exercise sessions and to nutrition and psychologist sessions

SECONDARY OUTCOMES:
Changes in (estimated) cardiorespiratory fitness | 3-6 months (from 1st treatment to surgery)
  Mile-time test
Changes in muscle strength | 3-6 months (from 1st treatment to surgery)
  Handgrip by dynamometry
Changes in body mass index | 3-6 months (from 1st treatment to surgery)
  BMI (Body Mass Index kg/sm)
Changes in body composition | 3-6 months (from 1st treatment to surgery)
  waist, hip, calf circumferences
Changes in levels of physical activity at week | 3-6 months (from 1st treatment to surgery)
  Accelerometry
Changes in quality of life | 3-6 months (from before1st treatment to surgery)
  EORTC-QLQ-C30 (European Organization for Research and Treatment of Cancer. Quality of Life questionnaire. C30. all scores of the QLQ-C30 were transformed linearly so that all scales ranged from 0 to 100. In the function scales higher scores represent a better level of functioning while in the case of symptom scales/items higher scores mark a higher level of symptomatology or problems.
Describe changes in fatigue levels | 3-6 months (from before 1st treatment to surgery)
  PERFORM (Multidimensional scale 12-60. The higher the less fatigue)
Dose intensity in neoadjuvant treatment | 3-6 months (from 1st treatment to surgery)
  percentage of intended doses that are administered in the due time
Describe post-surgical complications | three months
  Surgical wound and pancreatic fistula
Nutritional status | 3-6 months (from 1st treatment to surgery)
  body mass index
Percentage of pathological complete responses | 4-6 weeks after surgery
  Percentage of patients with no viable cells in the surgical specimen
Percentage of patients receiving adjuvant therapy | Three months after surgery
  Patients that received at least two cycles after surgery
Hindrances and facilitators of patients | During the prehabilitation program (3-6 months for each patient)
  Qualitative methods. semi-structured interviews and observation
Anxiety and depression | 3-6 months (from 1st treatment to surgery)
  Hospital Anxiety and Depression Scale questionnaire. Values 8-21. The higher the worse

OTHER OUTCOMES:
Circulating tumor DNA and mutational variations | before initiating chemotherapy
  circulant tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ruiz-Casado, MD, Principal Investigator — HU Puerta de Hierro Majadahonda
Locations (1):
- Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain

REFERENCES:
- [Background] Alejo LB, Pagola-Aldazabal I, Fiuza-Luces C, Huerga D, de Torres MV, Verdugo AS, Ortega Solano MJ, Felipe JL, Lucia A, Ruiz-Casado A. Exercise prehabilitation program for patients under neoadjuvant treatment for rectal cancer: A pilot study. J Cancer Res Ther. 2019 Jan-Mar;15(1):20-25. doi: 10.4103/jcrt.JCRT_30_17. PMID 30880749
- [Background] Ausania F, Senra P, Melendez R, Caballeiro R, Ouvina R, Casal-Nunez E. Prehabilitation in patients undergoing pancreaticoduodenectomy: a randomized controlled trial. Rev Esp Enferm Dig. 2019 Aug;111(8):603-608. doi: 10.17235/reed.2019.6182/2019. PMID 31232076
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Bolshinsky V, Li MH, Ismail H, Burbury K, Riedel B, Heriot A. Multimodal Prehabilitation Programs as a Bundle of Care in Gastrointestinal Cancer Surgery: A Systematic Review. Dis Colon Rectum. 2018 Jan;61(1):124-138. doi: 10.1097/DCR.0000000000000987. PMID 29219922
- [Background] Bundred JR, Kamarajah SK, Hammond JS, Wilson CH, Prentis J, Pandanaboyana S. Prehabilitation prior to surgery for pancreatic cancer: A systematic review. Pancreatology. 2020 Sep;20(6):1243-1250. doi: 10.1016/j.pan.2020.07.411. Epub 2020 Aug 3. PMID 32826168
- [Background] Carli F, Silver JK, Feldman LS, McKee A, Gilman S, Gillis C, Scheede-Bergdahl C, Gamsa A, Stout N, Hirsch B. Surgical Prehabilitation in Patients with Cancer: State-of-the-Science and Recommendations for Future Research from a Panel of Subject Matter Experts. Phys Med Rehabil Clin N Am. 2017 Feb;28(1):49-64. doi: 10.1016/j.pmr.2016.09.002. PMID 27913000
- [Background] Chandrabalan VV, McMillan DC, Carter R, Kinsella J, McKay CJ, Carter CR, Dickson EJ. Pre-operative cardiopulmonary exercise testing predicts adverse post-operative events and non-progression to adjuvant therapy after major pancreatic surgery. HPB (Oxford). 2013 Nov;15(11):899-907. doi: 10.1111/hpb.12060. Epub 2013 Feb 20. PMID 23458160
- [Background] Djarv T, Metcalfe C, Avery KN, Lagergren P, Blazeby JM. Prognostic value of changes in health-related quality of life scores during curative treatment for esophagogastric cancer. J Clin Oncol. 2010 Apr 1;28(10):1666-70. doi: 10.1200/JCO.2009.23.5143. Epub 2010 Mar 1. PMID 20194863
- [Background] Florez Bedoya CA, Cardoso ACF, Parker N, Ngo-Huang A, Petzel MQ, Kim MP, Fogelman D, Romero SG, Wang H, Park M, Katz MHG, Schadler KL. Exercise during preoperative therapy increases tumor vascularity in pancreatic tumor patients. Sci Rep. 2019 Sep 27;9(1):13966. doi: 10.1038/s41598-019-49582-3. PMID 31562341
- [Background] González-Cutre D, Sicilia A, Sierra AC et al. Understanding the need for novelty from the perspective of self-determination theory. Personality and Individual Differences 2016; 102:159-169
- [Background] Gruber ES, Jomrich G, Kaider A, Gnant M, Sahora K, Schindl M. The Prognostic Index Independently Predicts Survival in Patients with Pancreatic Ductal Adenocarcinoma Undergoing Resection. Ann Surg Oncol. 2020 Jun;27(6):2017-2024. doi: 10.1245/s10434-019-08161-6. Epub 2020 Jan 3. PMID 31900809
- [Background] Jie B, Jiang ZM, Nolan MT, Zhu SN, Yu K, Kondrup J. Impact of preoperative nutritional support on clinical outcome in abdominal surgical patients at nutritional risk. Nutrition. 2012 Oct;28(10):1022-7. doi: 10.1016/j.nut.2012.01.017. Epub 2012 Jun 5. PMID 22673593
- [Background] Jones LW, Peddle CJ, Eves ND, Haykowsky MJ, Courneya KS, Mackey JR, Joy AA, Kumar V, Winton TW, Reiman T. Effects of presurgical exercise training on cardiorespiratory fitness among patients undergoing thoracic surgery for malignant lung lesions. Cancer. 2007 Aug 1;110(3):590-8. doi: 10.1002/cncr.22830. PMID 17582629
- [Background] Jones LW, Eves ND, Haykowsky M, Joy AA, Douglas PS. Cardiorespiratory exercise testing in clinical oncology research: systematic review and practice recommendations. Lancet Oncol. 2008 Aug;9(8):757-65. doi: 10.1016/S1470-2045(08)70195-5. PMID 18672211
- [Background] Kodama S, Saito K, Tanaka S, Maki M, Yachi Y, Asumi M, Sugawara A, Totsuka K, Shimano H, Ohashi Y, Yamada N, Sone H. Cardiorespiratory fitness as a quantitative predictor of all-cause mortality and cardiovascular events in healthy men and women: a meta-analysis. JAMA. 2009 May 20;301(19):2024-35. doi: 10.1001/jama.2009.681. PMID 19454641
- [Background] Kokkinos P, Faselis C, Myers J, Sui X, Zhang J, Blair SN. Age-specific exercise capacity threshold for mortality risk assessment in male veterans. Circulation. 2014 Aug 19;130(8):653-8. doi: 10.1161/CIRCULATIONAHA.114.009666. Epub 2014 Jun 17. PMID 24938279
- [Background] Kurita Y, Kobayashi N, Tokuhisa M, Goto A, Kubota K, Endo I, Nakajima A, Ichikawa Y. Sarcopenia is a reliable prognostic factor in patients with advanced pancreatic cancer receiving FOLFIRINOX chemotherapy. Pancreatology. 2019 Jan;19(1):127-135. doi: 10.1016/j.pan.2018.11.001. Epub 2018 Nov 10. PMID 30473464
- [Background] Lee CHA, Kong JC, Ismail H, Riedel B, Heriot A. Systematic Review and Meta-analysis of Objective Assessment of Physical Fitness in Patients Undergoing Colorectal Cancer Surgery. Dis Colon Rectum. 2018 Mar;61(3):400-409. doi: 10.1097/DCR.0000000000001017. PMID 29377872
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Morielli AR, Usmani N, Boule NG, Severin D, Tankel K, Joseph K, Nijjar T, Fairchild A, Courneya KS. Feasibility, Safety, and Preliminary Efficacy of Exercise During and After Neoadjuvant Rectal Cancer Treatment: A Phase II Randomized Controlled Trial. Clin Colorectal Cancer. 2021 Sep;20(3):216-226. doi: 10.1016/j.clcc.2021.05.004. Epub 2021 May 26. PMID 34158253
- [Background] O'Connor D, Brown M, Eatock M, Turkington RC, Prue G. Exercise efficacy and prescription during treatment for pancreatic ductal adenocarcinoma: a systematic review. BMC Cancer. 2021 Jan 9;21(1):43. doi: 10.1186/s12885-020-07733-0. PMID 33422020
- [Background] Ross R, Blair SN, Arena R, Church TS, Despres JP, Franklin BA, Haskell WL, Kaminsky LA, Levine BD, Lavie CJ, Myers J, Niebauer J, Sallis R, Sawada SS, Sui X, Wisloff U; American Heart Association Physical Activity Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Cardiovascular and Stroke Nursing; Council on Functional Genomics and Translational Biology; Stroke Council. Importance of Assessing Cardiorespiratory Fitness in Clinical Practice: A Case for Fitness as a Clinical Vital Sign: A Scientific Statement From the American Heart Association. Circulation. 2016 Dec 13;134(24):e653-e699. doi: 10.1161/CIR.0000000000000461. Epub 2016 Nov 21. PMID 27881567
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Smith HR. Depression in cancer patients: Pathogenesis, implications and treatment (Review). Oncol Lett. 2015 Apr;9(4):1509-1514. doi: 10.3892/ol.2015.2944. Epub 2015 Feb 9. PMID 25788991
- [Background] Smith TB, Stonell C, Purkayastha S, Paraskevas P. Cardiopulmonary exercise testing as a risk assessment method in non cardio-pulmonary surgery: a systematic review. Anaesthesia. 2009 Aug;64(8):883-93. doi: 10.1111/j.1365-2044.2009.05983.x. PMID 19604193
- [Background] Spencer JC, Wheeler SB. A systematic review of Motivational Interviewing interventions in cancer patients and survivors. Patient Educ Couns. 2016 Jul;99(7):1099-1105. doi: 10.1016/j.pec.2016.02.003. Epub 2016 Feb 8. PMID 26879805
- [Background] Tew GA, Ayyash R, Durrand J, Danjoux GR. Clinical guideline and recommendations on pre-operative exercise training in patients awaiting major non-cardiac surgery. Anaesthesia. 2018 Jun;73(6):750-768. doi: 10.1111/anae.14177. Epub 2018 Jan 13. PMID 29330843
- [Background] Tsimopoulou I, Pasquali S, Howard R, Desai A, Gourevitch D, Tolosa I, Vohra R. Psychological Prehabilitation Before Cancer Surgery: A Systematic Review. Ann Surg Oncol. 2015 Dec;22(13):4117-23. doi: 10.1245/s10434-015-4550-z. Epub 2015 Apr 14. PMID 25869228